CLINICAL TRIAL: NCT07338968
Title: A Long-Term Follow-Up Study of Subjects Completing the AU-011-301 (CoMpass) Trial of Bel-sar for Early Choroidal Melanoma (Indeterminate Lesions/Small Choroidal Melanomas)
Brief Title: A Long-Term Follow-Up Study of Subjects Completing the AU-011-301(CoMpass) for Early Choroidal Melanoma
Acronym: CoMpass
Status: Not yet recruiting | Type: Observational
Sponsor: Aura Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: AU-011-403
Record Dates: First submitted 2025-11-21; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Choroidal Melanoma; Indeterminate Lesions
Keywords: Ocular Melanoma; Small Choroidal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — The intention is to collect data for an additional ~5 years (Post AU-011-301 participation)

SUMMARY:
AU-011-403 is a multicenter long-term follow-up safety and efficacy study of subjects with early CM who previously participated in the AU-011-301 Phase 3 trial. There are no required interventions or use of AU-011 (bel-sar) in this long-term follow-up study

DETAILED DESCRIPTION:
Informed consent will be obtained for each subject, preferably during their participation in the AU-011-301 trial and no more than approximately 6 months after their AU-011-301 End of Trial (EoT)/Early Termination (ET) visit. All subjects will be followed for an additional ~5 years (not including AU-011-301 participation). The AU-011-301 assigned subject numbering will continue to be used in this study. The AU-011-301 randomization (treatment received) will continue to be masked during this study until the completion of the AU-011-301 trial and database lock. The purpose of this long-term follow-up study is to learn about how safe and how well bel-sar works over time in people who previously participated in the AU-011-301 study. This will include collecting data from both people who received bel-sar and those who received the sham procedure.

The AU-011-403 study will collect data on:

Long-term safety will be measured by collecting information about any side effects (adverse events) or serious medical problems (serious adverse events) that may occur.

Long-term effectiveness of treatment in AU-011-301 will be measured by looking at any changes in subject's early CM and/or changes in vision over time.

Disease progression, including whether the early CM spreads to other parts of the body (metastasis).

Survival outcomes, including overall survival and disease-specific survival. Long-term quality of life (QoL) will be measured by using questionnaires (EORTC-QLQ-C30 and EORTC-QLQ-OPT30).

This study will help determine how long the effects of bel-sar last and whether any long-term risks or benefits appear after the initial treatment period.

The information collected may also help improve treatment options and strategies for future patients with early CM.

ELIGIBILITY:
Inclusion Criteria:

* Have received bel-sar or sham treatment in the Aura-sponsored clinical trial AU-011-301.
* Be willing and able to consent to the AU-011-403 study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have received bel-sar or sham treatment in the Aura-sponsored clinical trial AU-011-301. NCT NCT06007690
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2033-08-15 (Estimated); Study Completion 2033-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs)/serious AEs. | 5 years
  The AU-011-403 study is the long-term follow-up study of participants previously treated in AU-011-301.Long-term safety will be assessed by measuring the incidence of adverse events (AEs) and serious adverse events (SAEs) occurring during the follow-up period. AEs will be coded using the same Medical Dictionary for Regulatory Activities version used in AU-011-301 (MedDRA)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Aura Biosciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Aura Biosciences — http://www.aurabiosciences.com